CLINICAL TRIAL: NCT03122301
Title: Effects of Stellate Ganglion Block on Hot Flashes in Hispanic Women With Breast Cancer: A Pilot Randomized Sham-Controlled Trial
Brief Title: Effects of Stellate Ganglion Block on Hot Flashes in Hispanic Women With Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped due to inadequate enrollment.
Sponsor: Northwestern University (Other)
Collaborators: Indiana University (Other); University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, David Walega, Associate Professor of Anesthesiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STU00204093
Record Dates: First submitted 2017-04-18; First posted 2017-04-20 (Actual); Results first posted 2022-06-03 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-07

CONDITIONS: Hot Flashes; Hot Flushes; Vasomotor Symptoms
MeSH Terms: conditions — Hot Flashes | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivicaine (Active Comparator): Stellate Ganglion Block Injection with bupivicaine
  Interventions: Drug: Stellate Ganglion Block injection with bupivicaine
- Saline (Sham Comparator): Saline injection
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Stellate Ganglion Block injection with bupivicaine — A computer-generated 1:1 block randomization scheme will be used to assign participants to receive either a SGB with bupivacaine or a sham injection with saline. Randomization will be performed by the injectionist immediately before the injection procedure by opening an opaque envelope to reveal the participant number and group assignment printed on an index card.
  Other Names: Marcaine
  Arms: Bupivicaine
Drug: Saline — sham injection with saline
  Arms: Saline

SUMMARY:
Vasomotor symptoms (hot flashes, night sweats, VMS) affect up to 65% of breast cancer survivors and negatively impact their quality of life. VMS in Hispanic women are significantly more severe as compared to non-Hispanic Caucasian women. Few effective treatments for VMS are available, especially in the underserved Hispanic and Spanish-speaking populations which is problematic, as Hispanics will comprise 20% of the U.S. population by 2025. Stellate ganglion nerve block (SGB) with local anesthetic, previously performed for chronic pain indications, has shown promise as a potential treatment for menopausal women with VMS in previous clinical trials, but has not been investigated in Hispanic or Spanish-Speaking women with breast cancer in a controlled study.

DETAILED DESCRIPTION:
In this study, investigators aim to assess the effects of SGB on VMS, sympathetic nervous system activity, depression and sleep in Hispanic and Spanish-Speaking women with breast cancer on endocrine therapy who take tamoxifen, aromatase inhibitors (AIs) or SERMS, in a prospective, randomized, sham-controlled pilot study.

Project Hypothesis: The frequency and intensity of subjective and objective VMS will be significantly lower in women randomized to active SGB as compared to sham control.

Project Scope: Hispanic and Spanish-speaking women with breast cancer on tamoxifen, aromatase inhibitors or SERMs with moderate to severe VMS will be enrolled as participants in this study. Eligible women will be specifically recruited from the oncology practice of Dr. Cesar Santa Maria, as well as Northwestern Memorial Hospital and other Northwestern affiliates.

Specific Goals and Objectives:

Goal 1: Determine the effect of stellate ganglion blockade (SGB) for reducing subjective and objective VMS in Hispanic women with breast cancer on endocrine therapy as this population is known to have a greater severity of VMS and has been notoriously underserved and understudied in the U.S. and in clinical trials.

Goal 2: Evaluate the effect of SGB on the sympathetic nervous system over time to gain new knowledge on the physiologic mechanism of SGB effects on VMS.

Goal 3: Evaluate the effect of SGB on mood, sleep, and quality of life in women with breast cancer on tamoxifen, AIs, or SERMs.

Goal 4: Using the results of this pilot study, investigators plan to submit an R01 grant to the National Cancer Institute in 2017 for a larger scale study.

ELIGIBILITY:
Inclusion Criteria:

1. Hispanic or Spanish speaking women aged 30 to 70 years
2. 28 or more reported moderate-to-very severe hot flashes per week
3. a minimum of two weeks of VMS diary recording prior to SGB
4. current use of tamoxifen, aromatase inhibitors, or SERMs for a breast cancer indication for at last six months
5. willingness to undergo fluoroscopy-guided SGB or sham treatment.
6. if participant is on an SSRI,SNRI or membrane stabilizer (pregabalin, gabapentin, for example), it must be a stable, unchanged dose for previous 3 months

Exclusion Criteria:

1. conditions that preclude SGB or sham intervention (e.g., anatomic abnormalities of the anterior neck or cervical spine; goiter, cardiac/pulmonary compromise; acute illness/infection; coagulopathy or bleeding disorder; allergic reactions/contraindications to a local anesthetic or contrast dye); pregnancy 2. use of treatments in the past 2 months that can affect VMS (e.g., use of oral or transdermal HT or contraceptives,

-

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Walega, MD, MSCI, Principal Investigator — Northwestern University
Locations (1):
- Anesthesiology Pain Medicine Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bupivicaine | Saline
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivicaine | Saline | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Customized [Mean (Full Range); unit: years]
  Age | 48 | 36 | 42 [36 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 2
Baseline Hot Flashes [Mean (Standard Deviation); unit: Number of hot flashes/night] — Mean number of hot flashes per night for one month before treatment as reported by the study participant.
  Number of hot flashes/night | 1.3 (1.94) | 4.58 (2.78) | 2.94 (2.91)

OUTCOME MEASURES:

1. Primary Outcome: 2 Month Subject Reported Daily Hot Flashes (Mean)
Description: 2 month subject reported daily hot flashes measured from day 60 to day 90 after treatment (mean value).
Time Frame: 2 months after treatment
Measure: Mean (Standard Deviation); unit: Number of hot flashes/night
Arm/Group | Bupivicaine | Saline
Number analyzed (Participants) | 1 | 1
Number of hot flashes/night | .36 (.37) | 4.13 (2.5)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Bupivicaine | Saline
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
This study was terminated due to low enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/01/NCT03122301/Prot_SAP_000.pdf